CLINICAL TRIAL: NCT04745351
Title: A Phase 3 Randomized, Double-Blind, Placebo-Controlled, Parallel Group, Multicenter Study Evaluating the Efficacy and Safety of Remdesivir in Participants With Severely Reduced Kidney Function Who Are Hospitalized for COVID-19
Brief Title: Study to Evaluate the Efficacy and Safety of Remdesivir in Participants With Severely Reduced Kidney Function Who Are Hospitalized for Coronavirus Disease 2019 (COVID-19)
Acronym: REDPINE
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The study was terminated due to study enrollment feasibility. This decision is not based on efficacy or safety concerns.
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GS-US-540-5912; 2020-005416-22 (EudraCT Number); DOH-27-012022-4779 (Registry Identifier: South African Clinical Trials Register)
Expanded Access: NCT04323761 (Approved for marketing)
Record Dates: First submitted 2021-02-08; First posted 2021-02-09 (Actual); Results first posted 2023-05-12 (Actual); Last update posted 2023-05-12 (Actual); Status verified 2023-04

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — remdesivir; Standard of Care

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Remdesivir (RDV) (Experimental): Participants will receive continued Standard of Care (SOC) therapy together with RDV 200 mg on Day 1 followed by RDV 100 mg from Day 2 up to Day 5.
  Interventions: Drug: Remdesivir; Drug: Standard of Care
- Placebo (Placebo Comparator): Participants will receive continued SOC therapy together with RDV matching placebo on Day 1 followed by RDV matching placebo from Day 2 up to Day 5.
  Interventions: Drug: RDV Placebo; Drug: Standard of Care

INTERVENTIONS:
Drug: Remdesivir — Administered as Intravenous (IV) infusion once daily
  Other Names: GS-5734™; Veklury®
  Arms: Remdesivir (RDV)
Drug: RDV Placebo — Administered as IV saline once daily
  Arms: Placebo
Drug: Standard of Care — Standard of Care Treatment for COVID-19 Infection

SUMMARY:
The primary objective of this study is to evaluate whether remdesivir (RDV, GS-5734™) reduces the composite risk of death or invasive mechanical ventilation (IMV) through Day 29 in participants with severely reduced kidney function who are hospitalized for coronavirus disease 2019 (COVID-19).

ELIGIBILITY:
Key Inclusion Criteria:

* Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2) positive as determined by Polymerase Chain Reaction (PCR) or other commercially available or public health assay (eg, Nucleic Acid Amplification Test (NAAT) and antigen tests) in any respiratory specimen
* Hospitalized for COVID-19
* Weighing at least 40 kilograms (kg)
* Oxygen (O2) saturation ≤ 94% on room air or requiring O2 supplement or Radiographic evidence of pulmonary infiltrates for COVID-19
* Have either:

  * a) Severely reduced kidney function (estimated Glomerular Filtration Rate (eGFR) < 30 mL/min/1.73 m^2), including people with end-stage kidney disease (ESKD) requiring chronic dialysis
  * b) Ongoing acute kidney injury (AKI): defined as a 50% increase in serum creatinine (SCr) within a 48-hour period that is sustained (ie, requires confirmatory SCr) for ≥ 6 hours despite supportive care
* The interval between COVID-19 symptoms onset and randomization is no more than 10 days

Key Exclusion Criteria:

* Received any investigational drug, RDV, or other antiviral treatment for COVID-19
* Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) > 5 times the upper limit of normal
* Invasive mechanical ventilation, noninvasive mechanical ventilation, extracorporeal membrane oxygenation (ECMO), or renal replacement therapy (RRT) for acute kidney injury (AKI)
* Positive serum pregnancy test at screening for women of childbearing potential or currently breastfeeding
* Known hypersensitivity to the study drug, metabolites, or formulation sulfobutylether-beta-cyclodextrin (SBECD)

Note: Other protocol defined Inclusion/Exclusion criteria may apply

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 249 (Actual)
Dates: Start 2021-03-31 (Actual); Primary Completion 2022-04-20 (Actual); Study Completion 2022-05-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (63):
- United States (41):
  - St. Vincent's Health System, Birmingham, Alabama
  - UAB Hospital, Birmingham, Alabama
  - Pulmonary Associates of Mobile, P.C., Mobile, Alabama
  - St. Joseph Hospital Eureka, Eureka, California
  - Hoag Memorial Hospital Presbyterian, 16200 Sand Canyon Ave, Irvine, California
  - Hoag Memorial Hospital Presbyterian, Newport Beach, California
  - Sutter Medical Center Sacramento, Sacramento, California
  - Torrance Memorial Medical Center, Torrance, California
  - MedStar Health Research Institute, Washington D.C., District of Columbia
  - George Washington Medical Faculty Associates, Washington D.C., District of Columbia
  - North Florida/ South Georgia Veterans Health System, Gainesville, Florida
  - Mayo Clinic Florida, Jacksonville, Florida
  - Genesis Clinical Research, Tampa, Florida
  - Northwestern Medicine Central DuPage Hospital, Winfield, Illinois
  - Baptist Health Lexington, Lexington, Kentucky
  - Tulane Medical Center, 2000 Canal St., New Orleans, Louisiana
  - Tulane Medical Center, New Orleans, Louisiana
  - Wake Forest University Health Sciences, Bethesda, Maryland
  - Holy Cross Hospital, 19801 Observation Dr, Germantown, Maryland
  - Holy Cross Hospital, Silver Spring, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Newton-Wellesley Hospital, Newton, Massachusetts
  - St. Clair Nephrology Research, Grosse Pointe Woods, Michigan
  - G.V. (Sonny) Montgomery VAMC, Jackson, Michigan
  - Mayo Clinic Hospital, Rochester, Minnesota
  - Saint Michael's Medical Center, Newark, New Jersey
  - University of New Mexico Hospital, Albuquerque, New Mexico
  - New York - Presbyterian Hospital/Weill Cornell Medical Center, New York, New York
  - Stony Brook University Hospital, Stony Brook, New York
  - Jacobi Medical Center, The Bronx, New York
  - PMG Infectious Disease Consultants (administrative), Portland, Oregon
  - Temple University Hospital, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Houston Methodist Hospital, Houston, Texas
  - Memorial Hermann Hospital at TMC, Houston, Texas
  - VCU Health Medical Center, Richmond, Virginia
  - Providence Regional Medical Center Everett, Everett, Washington
  - Swedish Medical Center, Seattle, Washington
  - Providence Health Care, Spokane, Washington
  - Providence Health Care, 5633 N Lidgerwood, Spokane, Washington
  - MultiCare Good Samaritan Hospital, Tacoma, Washington
- Brazil (4):
  - Hospital e Maternidade Celso Pierro/ Sociedade Campineira de Educacao e Instrucao/ PUC Campinas, Campinas
  - Hospital Nossa Senhora das Gracas, Curitiba
  - Fundacao Faculdade Regional de Medicina de Sao Jose do Rio Preto, São José do Rio Preto
  - Hospital Alemao Oswaldo Cruz, São Paulo
- Portugal (5):
  - Centro Hospitalar Cova da Beira EPE, Covilha
  - Hospital Nélio Mendonça,, Funchal
  - Centro Hospitalar Lisboa Ocidental, Lisbon
  - Centro Hospitalar do Porto - Hospital de Santo Antonio, Odivelas
  - Centro Hospitalar de Vila Nova de Gaia, Vila Nova de Gaia
- South Africa (2):
  - George Regional Hospital, George
  - Mediclinic Vergelegen, Somerset West
- Spain (8):
  - Hospital Universitario Germans Trias I Pujol, Badalona
  - Hospital del Mar, Barcelona
  - Hospital Universitari de Bellvitge, Barcelona
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital General Universitario de Elche, Elche
  - Hospital Universitario 12 de Octubre, Madrid
  - Complejo Asistencial Universitario de Salamanca - H. Clinico, Salamanca
  - Hospital General Universitario de Valencia, Valencia
- United Kingdom (3):
  - Barts Health NHS Trust, The Royal London Hospital, London
  - Kings College Hospital, London
  - Imperial College Healthcare NHS Trust, London

IPD SHARING:
Plan to Share IPD: Yes
Qualified external researchers may request IPD for this study after study completion. For more information, please visit our website at https://www.gileadclinicaltrials.com/transparency-policy/
Supporting Information: Study Protocol, SAP
Time Frame: 18 months after study completion
Access Criteria: A secured external environment with username, password, and RSA code.
URL: https://www.gileadclinicaltrials.com/transparency-policy/

REFERENCES:
- [Derived] Sise ME, Santos JR, Goldman JD, Tuttle KR, Teixeira JP, Seibert AF, Koullias Y, Llewellyn J, Regan S, Zhao Y, Huang H, Hyland RH, Osinusi A, Winter H, Humeniuk R, Hulter HN, Gottlieb RL, Fusco DN, Birne R, Stancampiano FF, Libertin CR, Small CB, Plate M, McPhail MJ; REDPINE Investigators. Efficacy and Safety of Remdesivir in People With Impaired Kidney Function Hospitalized for COVID-19 Pneumonia: A Randomized Clinical Trial. Clin Infect Dis. 2024 Nov 22;79(5):1172-1181. doi: 10.1093/cid/ciae333. PMID 38913574
- [Derived] Grundeis F, Ansems K, Dahms K, Thieme V, Metzendorf MI, Skoetz N, Benstoem C, Mikolajewska A, Griesel M, Fichtner F, Stegemann M. Remdesivir for the treatment of COVID-19. Cochrane Database Syst Rev. 2023 Jan 25;1(1):CD014962. doi: 10.1002/14651858.CD014962.pub2. PMID 36695483
- See also: Gilead Clinical Trials Website — https://www.gileadclinicaltrials.com/study/?id=GS-US-540-5912

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in Brazil, Portugal, Spain, the United Kingdom, and the United States.
Pre-assignment Details: 258 participants were screened.
Groups:
- Remdesivir (RDV): Participants received continued Standard of Care (SOC) therapy together with RDV 200 mg intravenous (IV) infusion on Day 1 followed by RDV 100 mg IV infusion from Day 2 up to Day 5.
- Placebo: Participants received continued SOC therapy together with RDV matching placebo IV saline on Day 1 followed by RDV matching placebo IV saline from Day 2 up to Day 5.
Period: Overall Study
Arm/Group | Remdesivir (RDV) | Placebo
Started | 166 | 83
Completed | 95 | 50
Not Completed | 71 | 33
Not completed — Death | 51 | 25
Not completed — Lost to Follow-up | 9 | 3
Not completed — Randomized but Never Treated | 3 | 3
Not completed — Adverse Event | 4 | 0
Not completed — Withdrew Consent | 1 | 2
Not completed — Investigator's Discretion | 2 | 0
Not completed — Protocol Violation | 1 | 0

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set included all participants who were randomized into the study and had received at least 1 dose of study drug.
Groups:
- Remdesivir (RDV): Participants received continued SOC therapy together with RDV 200 mg IV infusion on Day 1 followed by RDV 100 mg IV infusion from Day 2 up to Day 5.
- Total: Total of all reporting groups
Arm/Group | Remdesivir (RDV) | Placebo | Total
Number analyzed (Participants) | 163 | 80 | 243
Age, Continuous [Mean (Standard Deviation); unit: years] | 68 (14.1) | 71 (13.0) | 69 (13.8)
Age, Customized [Count of Participants; unit: Participants]
  Age Categorical: < 18 Years | 0 | 0 | 0
  Age Categorical: >= 18 to < 65 Years | 70 | 22 | 92
  Age Categorical: >= 65 Years | 93 | 58 | 151
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 71 | 33 | 104
  Male | 92 | 47 | 139
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 23 | 8 | 31
  Not Hispanic or Latino | 135 | 72 | 207
  Unknown or Not Reported | 5 | 0 | 5
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: American Indian or Alaska Native | 1 | 0 | 1
  Race: Asian | 4 | 2 | 6
  Race: Black | 43 | 18 | 61
  Race: Native Hawaiian or Pacific Islander | 1 | 0 | 1
  Race: White | 104 | 55 | 159
  Race: Other | 8 | 3 | 11
  Race: Unknown or Not Reported | 2 | 2 | 4
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 121 | 59 | 180
  Spain | 26 | 13 | 39
  Portugal | 13 | 6 | 19
  United Kingdom | 2 | 2 | 4
  Brazil | 1 | 0 | 1
Clinical Status (8-point Ordinal Scale) [Count of Participants; unit: Participants] — The 8-point Ordinal scale assesses the clinical status of participants:1.Not hospitalized, no limitations on activities;2.Not hospitalized, limitation on activities/requiring home oxygen;3.Hospitalized,not requiring supplemental oxygen,no longer require ongoing medical care; 4.Hospitalized,not requiring supplemental oxygen-require ongoing medical care for COVID-19-specific medical care;5.Hospitalized,supplemental oxygen;6.Hospitalized,on noninvasive ventilation or highflow oxygen devices;7.Hospitalized,on invasive mechanical ventilation (IMV)/extracorporeal membrane oxygenation (ECMO);8.Death.
  Participants
    Score: 1 | 0 | 0 | 0
    Score: 2 | 0 | 0 | 0
    Score: 3 | 0 | 0 | 0
    Score: 4 | 36 | 18 | 54
    Score: 5 | 97 | 47 | 144
    Score: 6 | 30 | 15 | 45
    Score: 7 | 0 | 0 | 0
    Score: 8 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With All-cause Death or Invasive Mechanical Ventilation (IMV) Through Day 29
Description: This is the combined outcome measure reporting the percentage of participants with all-cause death or IMV through Day 29. The reported percentage was from the Kaplan-Meier estimate.
Time Frame: First dose date up to Day 29
Population: Full Analysis Set included all participants who were randomized into the study and had received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Remdesivir (RDV) | Placebo
Number analyzed (Participants) | 163 | 80
percentage of participants | 30.2 | 33.5
Statistical Analysis 1: Comparison: Remdesivir (RDV) vs Placebo; Test type: Superiority; p = 0.6132, Log Rank — P-value was calculated from stratified log-rank test, stratified by the baseline stratification factors; Hazard Ratio (HR) = 0.816, 95% CI 2-sided [0.504 to 1.321]

2. Secondary Outcome: All-cause Mortality Through Day 29
Description: The reported percentage was from the Kaplan-Meier estimate.
Time Frame: First dose date up to Day 29
Population: Participants in the Full Analysis Set were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Remdesivir (RDV) | Placebo
Number analyzed (Participants) | 163 | 80
percentage of participants | 25.9 | 29.7
Statistical Analysis 1: Comparison: Remdesivir (RDV) vs Placebo; Test type: Superiority; p = 0.3881, Log Rank — P-value was calculated from stratified log-rank test stratified by the baseline stratification factors; Hazard Ratio (HR) = 0.830, 95% CI 2-sided [0.497 to 1.388]

3. Secondary Outcome: Percentage of Participants With Initiation of IMV Through Day 29
Description: The reported percentage was the cumulative-incidence estimate.
Time Frame: First dose date up to Day 29
Population: Participants in the Full Analysis Set were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Remdesivir (RDV) | Placebo
Number analyzed (Participants) | 163 | 80
percentage of participants | 13.8 | 12.8
Statistical Analysis 1: Comparison: Remdesivir (RDV) vs Placebo; Test type: Superiority; p = 0.9116, Regression, Cox — The treatment effect p-value was calculated using Cox model with death as the competing risk and baseline stratification factors as covariates; Hazard Ratio (HR) = 1.043, 95% CI 2-sided [0.493 to 2.207]

4. Secondary Outcome: Time to Recovery Without Subsequent Worsening (Defined as an Ordinal Scale Score of > 4) by Day 29
Description: Time to recovery is the time from first dose to recovery. Recovery is defined as the first day on which the participant with a baseline score ≥ 4, satisfies categories 1, 2, or 3 from the 8-point ordinal scale: 1) Non-hospitalized, no limitations on activities; 2) Non-hospitalized, limitations on activities/requiring home oxygen; 3) Hospitalized, not requiring supplemental oxygen; 4) Hospitalized, not requiring supplemental oxygen - requiring ongoing medical care for COVID-19; 5) Hospitalized, supplemental oxygen; 6) Hospitalized, on noninvasive ventilation; 7) Hospitalized, on invasive mechanical ventilation or extracorporeal membrane oxygenation (ECMO); 8) Death. Cumulative incidence was reported.
Time Frame: First dose date up to Day 29
Population: Participants in the Full Analysis Set were analyzed.
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Remdesivir (RDV) | Placebo
Number analyzed (Participants) | 163 | 80
days | 20 [7 to NA] — Upper bound of range (Q3) was not estimable due to less than 75% of participants with recovery. | 19 [7 to NA] — Upper bound of range (Q3) was not estimable due to less than 75% of participants with recovery.

5. Secondary Outcome: Time to Recovery Independent of Further Worsening by Day 29
Description: Time to recovery is the time from first dose to recovery. Recovery is defined as the first day on which the participant with a baseline score ≥ 4, satisfies categories 1, 2, or 3 from the 8-point ordinal scale: 1) Non-hospitalized, no limitations on activities; 2) Non-hospitalized, limitations on activities/requiring home oxygen; 3) Hospitalized, not requiring supplemental oxygen; 4) Hospitalized, not requiring supplemental oxygen - requiring ongoing medical care for COVID-19; 5) Hospitalized, supplemental oxygen; 6) Hospitalized, on noninvasive ventilation; 7) Hospitalized, on invasive mechanical ventilation or ECMO; 8) Death. Cumulative incidence was reported.
Time Frame: First dose date up to Day 29
Population: Participants in the Full Analysis Set were analyzed.
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Remdesivir (RDV) | Placebo
Number analyzed (Participants) | 163 | 80
days | 10 [6 to NA] — Q3 was not estimable due to less than 75% of participants with recovery. | 13 [6 to NA] — Q3 was not estimable due to less than 75% of participants with recovery.

6. Secondary Outcome: Percentage of Participants Within Each Clinical Status Category as Assessed by an 8-Point Ordinal Scale on Day 15
Description: Clinical status is derived from death, hospital discharge, and the ordinal scale. Each day, the worst (highest) score from the previous day was recorded. The 8-point Ordinal scale is as follows: 1. Not hospitalized, no limitations on activities; 2. Not hospitalized, limitation on activities and/or requiring home oxygen; 3. Hospitalized, not requiring supplemental oxygen - no longer requires ongoing medical care (other than per-protocol RDV/saline as placebo administration); 4. Hospitalized, not requiring supplemental oxygen - requiring ongoing medical care for COVID-19-specific medical care (other than per-protocol RDV administration); 5. Hospitalized, supplemental oxygen; 6. Hospitalized, on noninvasive ventilation or high-flow oxygen devices; 7. Hospitalized, on IMV or ECMO; and 8. Death. Higher scores indicate worse clinical status.
Time Frame: Day 15
Population: Participants in the Full Analysis Set were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Remdesivir (RDV) | Placebo
Number analyzed (Participants) | 163 | 80
percentage of participants
  Score: 1 | 0 | 0
  Score: 2 | 48.5 | 48.8
  Score: 3 | 5.5 | 2.5
  Score: 4 | 9.2 | 7.5
  Score: 5 | 6.1 | 11.3
  Score: 6 | 8.0 | 5.0
  Score: 7 | 4.9 | 6.3
  Score: 8 | 17.8 | 18.8
Statistical Analysis 1: Comparison: Remdesivir (RDV) vs Placebo; Test type: Superiority; p = 0.8541, Proportional odds model — P-value was analysed from proportional odds model including treatment as the independent variable

7. Secondary Outcome: Percentage of Participants Within Each Clinical Status Category as Assessed by an 8-Point Ordinal Scale on Day 29
Description: as for outcome 6
Time Frame: Day 29
Population: Participants in the Full Analysis Set were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Remdesivir (RDV) | Placebo
Number analyzed (Participants) | 163 | 80
percentage of participants
  Score: 1 | 11.7 | 16.3
  Score: 2 | 42.9 | 45.0
  Score: 3 | 3.1 | 2.5
  Score: 4 | 4.3 | 1.3
  Score: 5 | 9.2 | 2.5
  Score: 6 | 1.8 | 1.3
  Score: 7 | 1.8 | 2.5
  Score: 8 | 25.2 | 28.8
Statistical Analysis 1: Comparison: Remdesivir (RDV) vs Placebo; Test type: Superiority; p = 0.4974, Proportional odds model — P-value was analysed from proportional odds model including treatment as the independent variable

8. Secondary Outcome: Renal Replacement Therapy (RRT)-Free Days (Among Those Without End-Stage Kidney Disease [ESKD] at Baseline) Through Day 29
Description: The number of RRT free days were calculated as the number of full days from Day 1 to Day 29 on which the participant was alive and did not receive RRT.
Time Frame: First dose date up to Day 29
Population: Participants without ESKD at baseline in the Full Analysis Set with available data were analyzed.
Measure: Median (Full Range); unit: days
Arm/Group | Remdesivir (RDV) | Placebo
Number analyzed (Participants) | 104 | 50
days | 29 [1 to 29] | 29 [4 to 29]
Statistical Analysis 1: Comparison: Remdesivir (RDV) vs Placebo; Test type: Superiority; p = 0.4283, Wilcoxon (Mann-Whitney) — P-value was calculated based on Wilcoxon rank sum test

9. Secondary Outcome: Percentage of Participants With Recovery Without Subsequent Worsening (Defined as an Ordinal Scale Score of > 4) Through Day 29
Description: Recovery is defined as the first day on which the participant with a baseline score >= 4, satisfies categories 1, 2, or 3 from the 8-point ordinal scale including: 1) Non-hospitalized, no limitations on activities; 2) Non-hospitalized, limitations on activities/requiring home oxygen; 3) Hospitalized, not requiring supplemental oxygen; 4) Hospitalized, not requiring supplemental oxygen - requiring ongoing medical care for COVID-19; 5) Hospitalized, supplemental oxygen; 6) Hospitalized, on noninvasive ventilation; 7) Hospitalized, on IMV or ECMO; 8) Death.
Time Frame: First dose date up to Day 29
Population: Participants in the Full Analysis Set were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Remdesivir (RDV) | Placebo
Number analyzed (Participants) | 163 | 80
percentage of participants | 57.7 | 63.8
Statistical Analysis 1: Comparison: Remdesivir (RDV) vs Placebo; Test type: Superiority; p = 0.2773, Cochran-Mantel-Haenszel — The treatment effect p-value was calculated using Cochran-Mantel-Haenszel (CMH) analysis including baseline stratification factors; Relative risk = 0.89, 95% CI 2-sided [0.731 to 1.091]

10. Secondary Outcome: Percentage of Participants With Recovery Independent of Further Worsening Through Day 29
Description: as for outcome 9
Time Frame: First dose date up to Day 29
Population: Participants in the Full Analysis Set were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Remdesivir (RDV) | Placebo
Number analyzed (Participants) | 163 | 80
percentage of participants | 66.3 | 67.5
Statistical Analysis 1: Comparison: Remdesivir (RDV) vs Placebo; Test type: Superiority; p = 0.7538, Cochran-Mantel-Haenszel — The treatment effect p-value was calculated using CMH analysis including baseline stratification factors; Relative risk = 0.97, 95% CI 2-sided [0.819 to 1.155]

11. Secondary Outcome: Percentage of Participants Experiencing Serious Adverse Events (SAEs)
Description: An SAE was defined as an event that, at any dose, results in the following: Death, a life-threatening situation, inpatient hospitalization or prolongation of existing hospitalization, persistent or significant disability/incapacity, a congenital anomaly/birth defect, a medically important event or reaction which may not be immediately life-threatening or result in death or hospitalization but may jeopardize the participant or may require intervention to prevent one of the other outcomes constituting SAEs.
Time Frame: First dose date up to last dose date (Maximum: 5 days) plus 30 days
Population: as for baseline characteristics
Measure: Number; unit: percentage of participants
Arm/Group | Remdesivir (RDV) | Placebo
Number analyzed (Participants) | 163 | 80
percentage of participants | 50.3 | 50.0

12. Secondary Outcome: Percentage of Participants Who Permanently Discontinued Investigational Drug Due to Adverse Events (AEs)
Description: An AE is any untoward medical occurrence in a clinical study participant administered an investigational drug, which does not necessarily have a causal relationship with the treatment. An AE can therefore be any unfavorable and/or unintended sign, symptom, or disease temporally associated with the use of an investigational drug, whether or not the AE is considered related to the investigational drug.
Time Frame: First dose date up to last dose date (Maximum: 5 days)
Population: Participants in the Safety Analysis Set were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Remdesivir (RDV) | Placebo
Number analyzed (Participants) | 163 | 80
percentage of participants | 4.9 | 1.3

ADVERSE EVENTS:
Time Frame: All-Cause Mortality: Randomization up to last follow-up visit (maximum of 15 weeks); Adverse Events: First dose date up to last dose date (maximum: 5 days) plus 30 days
Description: All-Cause Mortality: All Randomized Analysis Set included all participants who were randomized in the study.
  Adverse Events: Safety Analysis Set included all participants who were randomized into the study and had received at least 1 dose of study drug.
Arm/Group | Remdesivir (RDV) | Placebo
All-Cause Mortality (participants affected / at risk) | 55/166 | 26/83
Serious Adverse Events (participants affected / at risk) | 82/163 | 40/80
Other Adverse Events (participants affected / at risk) | 60/163 | 34/80
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Remdesivir (RDV) (N=163) | Placebo (N=80)
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Pancytopenia (Blood and lymphatic system disorders) | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 3 | 0
Atrial flutter (Cardiac disorders) | 1 | 0
Atrioventricular block (Cardiac disorders) | 1 | 0
Bradycardia (Cardiac disorders) | 2 | 0
Cardiac arrest (Cardiac disorders) | 8 | 1
Cardiac failure (Cardiac disorders) | 2 | 0
Cardiac failure acute (Cardiac disorders) | 2 | 1
Cardiac failure congestive (Cardiac disorders) | 2 | 0
Cardiac ventricular thrombosis (Cardiac disorders) | 0 | 1
Cardio-respiratory arrest (Cardiac disorders) | 2 | 3
Cardiogenic shock (Cardiac disorders) | 1 | 0
Pulseless electrical activity (Cardiac disorders) | 3 | 0
Supraventricular tachycardia (Cardiac disorders) | 2 | 0
Ventricular tachycardia (Cardiac disorders) | 1 | 0
Adrenal insufficiency (Endocrine disorders) | 1 | 0
Duodenal perforation (Gastrointestinal disorders) | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 | 1
Intestinal perforation (Gastrointestinal disorders) | 1 | 0
Large intestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 2 | 0
Death (General disorders) | 1 | 0
General physical health deterioration (General disorders) | 1 | 0
Multiple organ dysfunction syndrome (General disorders) | 4 | 1
Pyrexia (General disorders) | 1 | 0
Sudden death (General disorders) | 1 | 0
Hepatic ischaemia (Hepatobiliary disorders) | 1 | 0
Aspergillus infection (Infections and infestations) | 1 | 0
Bacteraemia (Infections and infestations) | 3 | 0
Bacteroides bacteraemia (Infections and infestations) | 0 | 1
Bronchopulmonary aspergillosis (Infections and infestations) | 1 | 0
Covid-19 (Infections and infestations) | 2 | 3
Covid-19 pneumonia (Infections and infestations) | 3 | 1
Cystitis (Infections and infestations) | 1 | 0
Cytomegalovirus infection reactivation (Infections and infestations) | 1 | 1
Device related bacteraemia (Infections and infestations) | 0 | 1
Endocarditis bacterial (Infections and infestations) | 1 | 0
Gangrene (Infections and infestations) | 0 | 1
Peritonitis (Infections and infestations) | 1 | 0
Pneumocystis jirovecii infection (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 2 | 0
Pneumonia bacterial (Infections and infestations) | 2 | 1
Postoperative abscess (Infections and infestations) | 0 | 1
Pulmonary sepsis (Infections and infestations) | 1 | 0
Pyelonephritis acute (Infections and infestations) | 2 | 0
Respiratory tract infection (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 5 | 2
Septic shock (Infections and infestations) | 6 | 2
Superinfection bacterial (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0
Dialysis related complication (Injury, poisoning and procedural complications) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 2 | 0
Subdural haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Wound haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Glomerular filtration rate abnormal (Investigations) | 0 | 1
Lipase increased (Investigations) | 1 | 0
Acidosis (Metabolism and nutrition disorders) | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 2
Hyperlipasaemia (Metabolism and nutrition disorders) | 1 | 0
Hypervolaemia (Metabolism and nutrition disorders) | 0 | 1
Lactic acidosis (Metabolism and nutrition disorders) | 1 | 0
Metabolic acidosis (Metabolism and nutrition disorders) | 1 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Dementia (Nervous system disorders) | 1 | 0
Depressed level of consciousness (Nervous system disorders) | 2 | 0
Ischaemic stroke (Nervous system disorders) | 1 | 0
Metabolic encephalopathy (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 1 | 0
Delirium (Psychiatric disorders) | 1 | 0
Mental status changes (Psychiatric disorders) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 5 | 1
End stage renal disease (Renal and urinary disorders) | 0 | 1
Renal impairment (Renal and urinary disorders) | 0 | 1
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 10 | 4
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 6 | 2
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumomediastinum (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory acidosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 7 | 10
Aortic stenosis (Vascular disorders) | 0 | 1
Hypertension (Vascular disorders) | 0 | 1
Hypertensive urgency (Vascular disorders) | 0 | 1
Hypotension (Vascular disorders) | 7 | 0
Malignant hypertension (Vascular disorders) | 1 | 0
Peripheral arterial occlusive disease (Vascular disorders) | 0 | 1
Shock (Vascular disorders) | 2 | 0
Shock haemorrhagic (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Remdesivir (RDV) (N=163) | Placebo (N=80)
Anaemia (Blood and lymphatic system disorders) | 10 | 1
Atrial fibrillation (Cardiac disorders) | 7 | 4
Constipation (Gastrointestinal disorders) | 12 | 7
Nausea (Gastrointestinal disorders) | 12 | 3
Hyperglycaemia (Metabolism and nutrition disorders) | 7 | 5
Hyperkalaemia (Metabolism and nutrition disorders) | 13 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 8 | 4
Hypokalaemia (Metabolism and nutrition disorders) | 5 | 7
Hypomagnesaemia (Metabolism and nutrition disorders) | 3 | 4
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 4
Headache (Nervous system disorders) | 3 | 4
Agitation (Psychiatric disorders) | 5 | 4
Anxiety (Psychiatric disorders) | 5 | 7
Hypertension (Vascular disorders) | 4 | 6
Hypotension (Vascular disorders) | 12 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years.

DOCUMENTS (2):
  • Study Protocol (2021-08-27): https://cdn.clinicaltrials.gov/large-docs/51/NCT04745351/Prot_000.pdf
  • Statistical Analysis Plan (2022-07-22): https://cdn.clinicaltrials.gov/large-docs/51/NCT04745351/SAP_001.pdf